CLINICAL TRIAL: NCT04022707
Title: The Impact of Circuit Resistance Training on Cognition and Estimated Maximal Oxygen Consumption in Older Adults.
Brief Title: High Speed Circuit Training and Cognition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Joseph Signorile, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20190518
Record Dates: First submitted 2019-07-10; First posted 2019-07-17 (Actual); Last update posted 2020-05-18 (Actual); Status verified 2020-05

CONDITIONS: Educational Control; Resistance Training
Keywords: Elderly; Circuit training; Cognitive ability; Cardiovascular condition

STUDY DESIGN:
Intervention Model Description: Comparison of High-Speed Resistance training and educational control
Who Masked: Investigator, Outcomes Assessor
Masking Description: Tests will not be performed by the investigators providing the interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-Velocity Resistance Circuttraining (HVRCT) (Experimental): The participants will perform three circuits of 11 exercises that target the upper and lower body. Training will gradually increase over the first three weeks from 1 to 3 circuits.
  Interventions: Other: High-speed circuit resistance training; Other: Educational control
- Educational Control (CON) (Experimental): A supervised program will be provided to the participants that includes lectures on health and fitness.
  Interventions: Other: High-speed circuit resistance training; Other: Educational control

INTERVENTIONS:
Other: High-speed circuit resistance training — The program will include three circuits of 11 exercises that target the upper and lower body. Training will gradually increase over the first three week from 1 to 3 circuits.
  Other Names: High-velocity circuit training
Other: Educational control — Lectures on health and fitness
  Other Names: Control

SUMMARY:
The purpose of this research study is to see if a weight training program can make a positive change in participant fitness as measured by the ability to use oxygen and help the participant remember things.

DETAILED DESCRIPTION:
The purpose of this research study is to see if a weight training program can make a positive change in cardiac fitness, that is a person's ability to use oxygen; and, if the program can help a person's memory, as measured by some standard tests. The researchers will also ask the participant to attend two sessions with researchers at the Bascom-Palmer Eye Institute so they can take pictures of the participants' eyes to see how training changes the number of blood vessels. This can be used by doctors and other clinicians to evaluate improvements blood flow to the brain due to training.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women between 60 and 85 years of age (inclusive)
2. Ability to provide informed consent
3. No medical contraindication to participation in an exercise program including unstable or active untreated major medical illness (i.e., cardiovascular disease, neurological or neuromuscular diseases, stroke, cancer, etc.).

Exclusion Criteria:

1. Existing muscle-skeletal injury
2. Mini-mental score <18
3. Enrolled in another exercise program
4. Unstable or active major medical illness
5. Answer "Yes" to any questions on the Elder PAR-Q
6. Pregnancy

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Changes in Cognition due to training | Baseline, Week 14
  The MoCA will be used to detect mild cognitive impairment in the participants. The total possible score is 30 points; a score of 26 or above is considered normal.
Submaximal cycle ergometer test to measure aerobic capacity | Baseline, Week 14
  The Young Men's Club of America (YMCA) cycle ergometer test will be used to compute aerobic capacity using heart rate(HR). Predicted oxygen consumption will be computed using the HR of the last two consecutive workloads performed and the maximum workload. A maximal oxygen consumption of 36 milliliters per kilogram body weight per minute and above is considered excellent for men, while 30 milliliters per kilogram body weight per minute is considered excellent for women.
Change in episodic memory | Baseline, Week 14
  The National Institutes of Health (NIH) Toolbox: Picture Sequence Memory Test measures episodic memory. Participants are asked to reproduce a sequence of pictures that is shown on the screen. Participants are given credit for each adjacent pair of pictures they correctly place (i.e., if pictures in locations 7 and 8 are placed in that order and adjacent to each other anywhere, such as slots 1 and 2, one point is awarded), up to the maximum value for the sequence, which is one less than the sequence length or 17.
Change in attention and inhibitory control | Baseline, Week 14
  The NIH Toolbox Flanker test measures attention and inhibitory control. Participant focuses on a given stimulus while inhibiting attention to stimuli flanking it. This computed score ranges from 0-10, but if the score is less than 4, it indicates that the participant did not score high enough in accuracy (80 percent correct or less) to receive a reaction time score.
Change in working memory | Baseline, Week 14
  The NIH Toolbox List Sorting test measures working memory. Participant recalls and sequences different visually and orally presented stimuli. List Sorting is scored by summing the total number of items correctly recalled and sequenced on 1-List and 2-List, which can range from 0-26.
Change in speed of cognitive processing | Baseline, Week 14
  The NIH Toolbox Pattern Comparison Processing Speed test measures speed of processing. Participants discern whether two side-by-side pictures are the same or not, with 85 seconds to respond to as many items as possible. Items are simple so as to purely measure processing speed. The participant's raw score is the number of items answered correctly in 85 seconds of response time, with a range of 0-130.
Changes in the power muscles can produce | Baseline, Week 14
  The participants will stand up and down 3 times with a thin string attached to the participant's belt. A total of five attempts will be performed by each participant, and the highest power output will be selected for use in the analysis.
Change in retinal microvascular density as a marker of cortical changes | Baseline, Week 14
  Retinal microvascular density will be assessed using the Retinal Function Imager (RFI) scan protocol and Optical Coherence Tomography Angiography (OCTA). Pictures will be taken of the subject's retina as they look into a special self-contained camera system.

SECONDARY OUTCOMES:
Changes in body fat-free mass | Baseline, Week 14
  Fat-free mass will be measured using a Tanita BC-418 bioelectrical impedance scale.
Changes in body weight | Baseline, Week 14
  Body weight will be measured on an electronic scale

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Signorile, PhD, Principal Investigator — University of Miami
Locations (2):
- United States (2):
  - Max Orovitz Laboratories, Coral Gables, Florida
  - Laboratory of Neruomuscular Research and Active Aging, Coral Gables, Florida

IPD SHARING:
Plan to Share IPD: No